CLINICAL TRIAL: NCT06374121
Title: A Single-center, Pilot, Prospective, Randomized Clinical Study of Hypothermic Oxygenated Perfusion With or Without Adsorption in Histologically Evaluated Kidneys Retrieved From Marginal Donors
Brief Title: Kidney Perfusion With or Without Absorption
Acronym: POWER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POWER
Record Dates: First submitted 2024-04-10; First posted 2024-04-18 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Kidney Replacement
Keywords: Kidney perfusion; Absorption; Marginal donors

STUDY DESIGN:
Intervention Model Description: To compare the biochemical profiles of the perfusate obtained from 5 kidneys treated with perfusion and concomitant adsorption, with that of the perfusate obtained from 5 kidneys treated with perfusion without adsorption.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perfusion and concomitant adsorption (Experimental): Kidneys eligible for perfusion will be treated with the PerLife PerKidney system. Kidneys allocated to the adsorption subgroup will receive concomitant treatment with PerSorb cartridge.
  Interventions: Device: PerSorb cartridge (CytoSorbents Europe GmbH, Germany); Device: PerLife PerKidney
- Perfusion alone (Active Comparator): Kidneys eligible here will only be treated with the PerLife PerKidney system.
  Interventions: Device: PerLife PerKidney

INTERVENTIONS:
Device: PerSorb cartridge (CytoSorbents Europe GmbH, Germany) — This is a highly bio-/hemo-compatible, low-flow resistance polymer cartridge able to remove cytokines and other inflammatory mediators via adsorption.
  Arms: Perfusion and concomitant adsorption
Device: PerLife PerKidney — The system for ex vivo kidney reconditioning (Aferetica, Italy), which allows hypothermic oxygenated pulsatile perfusion of the organ.

SUMMARY:
In this single-center, pilot, prospective, randomized study, the investigators will compare the biochemical profiles of the perfusate and the functional parameters of five kidneys perfused with Integrated PerLife® system and "PerSorb ECOS-300CY ™" sorbent (adsorption groups) with the profiles of the perfusate and functional parameters of five matched kidneys perfused with Integrated PerLife® system only (non-adsorption group). Kidneys from marginal donors with a clinical indication to pre-transplant histological evaluation (donor >70-years-old or aged 60 to 69 years but with hypertension, diabetes and/or clinical proteinuria) will be allocated to perfusion with or without adsorption using a 1:1 randomization ratio. When both donor kidneys will have a score from 0 to 4, the two kidneys will be used for two single transplants. When one kidney will have a score from 0 to 4 and the other kidney will have a score of 5 or more, and when both kidneys will have a score from 5 to 7, the two kidneys will be transplanted together into the same recipient. If one kidney will have a score from 5 to 7 and the other kidney will have a score of 8 or greater, the two kidneys will be discarded. With the use of the minimization method, the randomization will be planned in order to have the same number of single or dual transplants in the perfusion kidney groups with or without adsorption. Donor selection, kidney evaluation and allocation and recipient management will be based on per center practice.

DETAILED DESCRIPTION:
In recent years, growing interest has been addressed to the use of dynamic preservation of the kidneys as a tool to improve graft function and survival. Retrospective analyses and a randomized controlled trial showed that pre-transplant machine perfusion (MP) is associated with a lower incidence of delayed graft function (DGF) and improved one-year graft survival as compared with static cold storage. However, the overall beneficial effect of MP on transplant outcomes is largely driven by treatment effect in recipients of grafts from marginal donors.

Hypothermic oxygenated perfusion has been found to reduce early allograft injury and to improve post-transplant outcomes in a randomized controlled trial of liver transplantation from older donors. In vitro studies show that perfusion reduces endothelial damage to the sinusoidal capillaries and increases adenosine triphosphate production. As far as kidney transplantation is concerned, little data is available on the outcomes of grafts treated with perfusion. In rat models of allogeneic kidney transplant, perfusion-treated grafts displayed better short-term function, less tubular injury, fewer interstitial infiltrates of immune cells and milder endothelial activation than the untreated counterparts.

MP is not only beneficial per se. It can also be exploited as a means to deliver additional treatment to the graft. For instance, there is in vivo evidence that hemoadsorption improves renal blood flow during perfusion and reduces the release of cytokines and prostaglandins at reperfusion in a porcine model of kidney transplantation. Beneficial effects of hemoadsorption have been documented in the setting of continuous renal replacement treatment for septic shock. In the setting of pre-transplant organ conditioning, cytokine adsorption paired to normothermic perfusion has been found to reduce inflammatory gene expression and increase oxidative phosphorylation pathway gene expression in human kidneys. Whether adsorption paired to perfusion reduces the inflammatory response and whether this is of clinical relevance in transplantation of histologically evaluated kidneys from marginal donors, is worth investigating.

ELIGIBILITY:
Inclusion Criteria:

* Males and females older than 50 years eligible for single or dual kidney transplant from marginal donors identified according to the NITp criteria (>70-year-old or 60 to 70 years with hypertension and/or diabetes and/or clinical proteinuria)
* Pre-transplant histological evaluation
* Histological score ≤ 7
* Written informed consent.

Exclusion Criteria:

* Any factor that represents a contraindication to receive a deceased donor kidney transplant according to the NITp criteria,
* Need for specific desensitization protocols because of a high immunological risk according to the NITp criteria,
* Active enrollment in concomitant intervention studies,
* Macroscopic vascular abnormalities that preclude the possibility of machine perfusion.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Oxidative stress markers | Every 30 minutes during clinical perfusion
  Glutathione S-transferase (GST), lactate dehydrogenase (LDH) and free lactate
Acute kidney injury markers | Every 30 minutes during clinical perfusion
  Neutrophil gelatinase-associated lipocalin (NGAL), kidney injury molecule-1 (KIM-1) and endothelin
Inflammatory cytokine markers | Every 30 minutes during clinical perfusion
  Interleukin-6 (IL-6), interleukin-10 (IL-10) and tumor necrosis factor alpha (TNF-⍺)
Complement activation markers | Every 30 minutes during clinical perfusion
  Complement factor 3a (C3a), complement factor 5a (C5a) and soluble membrane attack complex (sC5bC9)
Vascular resistances | Every 30 minutes during clinical perfusion
  Renal vascular resistances will be automatically collected through clinical perfuzione
Perfusate sample collection | At clinical perfusion start, after 1 hour, then after 4 hours from start and every 2 hours thereafter, up to perfusion end
  Pseudo-urine ureteral output will be separately assessed at sequential times during clinical perfusion

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Remuzzi, MD, Study Chair — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (1):
- ASST - Papa Giovanni XXIII - U.O. Nefrologia e Dialisi/ Mario Negri Institute for Pharmacological Research - Clinical Research Center for Rare Diseases Aldo e Cele Daccò, Bergamo, BG, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Remuzzi G, Grinyo J, Ruggenenti P, Beatini M, Cole EH, Milford EL, Brenner BM. Early experience with dual kidney transplantation in adults using expanded donor criteria. Double Kidney Transplant Group (DKG). J Am Soc Nephrol. 1999 Dec;10(12):2591-8. doi: 10.1681/ASN.V10122591. PMID 10589699
- [Background] Hosgood SA, Moore T, Kleverlaan T, Adams T, Nicholson ML. Haemoadsorption reduces the inflammatory response and improves blood flow during ex vivo renal perfusion in an experimental model. J Transl Med. 2017 Oct 25;15(1):216. doi: 10.1186/s12967-017-1314-5. PMID 29070045
- [Background] Brouwer WP, Duran S, Kuijper M, Ince C. Hemoadsorption with CytoSorb shows a decreased observed versus expected 28-day all-cause mortality in ICU patients with septic shock: a propensity-score-weighted retrospective study. Crit Care. 2019 Sep 18;23(1):317. doi: 10.1186/s13054-019-2588-1. PMID 31533846
- [Background] Hosgood SA, Hoff M, Nicholson ML. Treatment of transplant kidneys during machine perfusion. Transpl Int. 2021 Feb;34(2):224-232. doi: 10.1111/tri.13751. Epub 2020 Oct 19. PMID 32970886
- [Background] Ferdinand JR, Hosgood SA, Moore T, Ferro A, Ward CJ, Castro-Dopico T, Nicholson ML, Clatworthy MR. Cytokine absorption during human kidney perfusion reduces delayed graft function-associated inflammatory gene signature. Am J Transplant. 2021 Jun;21(6):2188-2199. doi: 10.1111/ajt.16371. Epub 2020 Nov 22. PMID 33098231